CLINICAL TRIAL: NCT04887025
Title: Exploratory Study of a Novel Oncolytic Vaccinia Virus Expressing Bispecific Antibody in the Treatment of Refractory/Relapsed B-cell Lymphoma
Brief Title: Exploratory Study of a Novel Oncolytic Vaccinia Virus RGV004 in the Treatment of Refractory/Relapsed B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Rongu Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2021002042
Record Dates: First submitted 2021-05-06; First posted 2021-05-14 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Relapsed or Refractory B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Subjects will be treated with RGV004 as a single injection, one time.
  Interventions: Biological: RGV004

INTERVENTIONS:
Biological: RGV004 — a genetically-engineered vaccinia virus (encoding CD19/CD3 bispecific antibody)

SUMMARY:
This is a dose-escalation, single-arm, single-center open study which aims to evaluate the maximum tolerated dose (MTD) and dose-dependent toxicity (DLT) of a novel oncolytic vaccinia virus expressing bispecific antibody RGV004 in patients with relapsed/refractory B-cell lymphoma,

DETAILED DESCRIPTION:
Oncolytic vaccinia virus administered by intratumoral injection

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, the upper limit is 75 years old, there is no restriction on men and women;
2. ECOG score 0-1;
3. Histological diagnosis of non-Hodgkin B-cell lymphoma (NHL) [diagnostic criteria according to WHO2008], including diffuse large B-cell lymphoma (DLBCL) non-specific, primary mediastinal large B-cell lymphoma (PMBCL) , Mantle cell lymphoma (MCL), transformed follicles Cell lymphoma (TFL) and other indolent B-cell NHL transformants;
4. CD19 positive (immunohistochemistry or flow cytometry);
5. DLBCL refractory (refractory) or relapse is defined as: complete remission is not achieved after 2-line treatment; disease appears during any treatment Disease progression, or disease stable time equal to or less than 6 months; or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation;
6. MCL: Complete remission has not been achieved after 2-line treatment (including BTK inhibitors); disease progression during any treatment, or disease stable time equal to or less than 6 months; or within 12 months after autologous hematopoietic stem cell transplantation Disease progression or recurrence;
7. There is at least one measurable superficial lesion, and any long diameter of the lymph node lesion is greater than 1.5 cm or any long diameter of the extranodal lesion is greater than 1.0 cm, and the PET-CT scan lesion is ingested (SUV is greater than the liver blood pool);
8. Peripheral blood neutrophil absolute value ≥ 2000/mm3, platelet ≥ 50,000/mm3;
9. Heart, liver and kidney functions: creatinine <1.5mg/dL; ALT (alanine aminotransferase) / AST (aspartate aminotransferase) below 2.5 times the upper limit of normal; total bilirubin <1.5mg/dL; cardiac ejection fraction ( EF) ≥50%;
10. Have sufficient understanding and voluntarily sign the informed consent form;
11. Women with fertility must undergo a negative serum pregnancy test and agree to implement effective birth control measures during the treatment phase and within 60 days after the last application of the oncolytic virus;
12. Male patients must agree to implement effective birth control measures during the study period and within 60 days after the last viral treatment.

Exclusion Criteria:

1. There is a history of other tumors;
2. Inoculate vaccinia vaccine 3 months before the study treatment and during the study treatment period;
3. Have received gene therapy or any type of oncolytic virus therapy within 3 months before the study treatment;
4. Other open wounds;
5. Active autoimmune diseases;
6. Active infection that cannot be controlled;
7. HIV infection, uncontrolled HBV, HCV, and syphilis infection;
8. Known lymphoma of the central nervous system;
9. Clinically important heart disease;
10. Allergic to albumin or egg products;
11. Have undergone similar operations such as organ transplantation;
12. Systemic treatment of skin diseases is required;
13. A history of severe systemic reactions or side effects after vaccinia vaccine injection;
14. Known dependence on alcohol or viruses;
15. Pregnant or lactating female patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
To define the Max tolerated dose (MTD) of RGV004 | Up to 28 days
  According to the principle of '3+3' dose escalation, if one patient experiences a Dose limiting Toxicity (DLT), up to three additional patients will be treated at the same dose level. If DLT is observed in only one of six patients treated at a given dose level, the next cohort of three patients will be treated at the next higher dose level. If two or more patients experience DLT at a particular dose level, then the dose escalation will cease and any subsequent patients will be treated at a lower dose level. Thus finding the Max tolerated dose (MTD)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 2 years
  To evaluate the number of Grade III and above side effects assessed by CTCAE v5.0 for patients who received intratumoral administration of RGV004 injection in patients with R/R B-cell lymphoma.

SECONDARY OUTCOMES:
Objective remission rate (ORR) | Up to 2 years
  The percentage of participants who achieved complete remission (CR) and partial remission (PR) over all participants
RGV004 viral DNA in blood | Up to 2 years
  Viral DNA load will be summarized by cohort
RGV004 viral shedding in saliva | Up to 2 years
  Viral DNA will be analyzed by qPCR
RGV004 viral shedding in urine | Up to 2 years
  Viral DNA will be analyzed by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No